CLINICAL TRIAL: NCT01326299
Title: Post Prandial Glucose Control Proof-of-Principle
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Director Clinical Research Operations, Abbott Nutrition
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BK92
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Nutritional ingredient (Active Comparator): Dissolve in water and consume with meal
  Interventions: Other: Nutritional ingredient
- Carbohydrate (Placebo Comparator): dissolve in water and consume with meal
  Interventions: Other: Carbohydrate placebo
- #1 Nutrtitional ingredient + Fiber (Experimental): Dissolve in water and consume with meal
  Interventions: Other: #1 Nutritional ingredient +Fiber
- #2 Nutritional ingredient + Fiber (Experimental): Dissolve in water and consume with meal
  Interventions: Other: #2 Nutritional ingredient + Fiber
- #3 Nutritional ingredient + Fiber (Experimental): Dissolve in water and consume with meal
  Interventions: Other: #3 Nutritional ingredient + Fiber

INTERVENTIONS:
Other: Carbohydrate placebo — dissolve in water and consume with meal
  Arms: Carbohydrate
Other: Nutritional ingredient — Dissolve in water and consume with meals
  Arms: Nutritional ingredient
Other: #1 Nutritional ingredient +Fiber — Dissolve in water and consume with meal
  Arms: #1 Nutrtitional ingredient + Fiber
Other: #2 Nutritional ingredient + Fiber — Dissolve in water and consume with meal
  Arms: #2 Nutritional ingredient + Fiber
Other: #3 Nutritional ingredient + Fiber — Dissolve in water and consume with meal
  Arms: #3 Nutritional ingredient + Fiber

SUMMARY:
The purpose of this study is to compare the postprandial glycemic response of subjects with type 2 diabetes when consuming a meal along with beverages containing various combinations of nutritional ingredients and fibers versus control beverage.

ELIGIBILITY:
Inclusion Criteria:

1. type 2 diabetes
2. between 21 and 75 years of age
3. male or a non-pregnant, non-lactating female, at least 6 weeks postpartum or postmenopausal or surgically sterile
4. BMI is > 18.5 kg/m2 and <35 kg/m2
5. HbA1c < 9.0%

Exclusion Criteria:

1. Subject uses exogenous insulin, exenatide, or sitagliptin phosphate
2. type 1 diabetes.
3. history of diabetic ketoacidosis.
4. current infection
5. active malignancy
6. has had a significant cardiovascular event or history of congestive heart failure.
7. end-stage organ failure or post organ transplant.
8. history of renal disease.
9. hepatic disease.
10. history of gastrointestinal disorders
11. chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV.
12. taking any herbals, dietary supplements, or medications, other than oral hypoglycemic medications
13. clotting or bleeding disorders.
14. allergic or intolerant to any ingredient found in the study products.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Positive AUC from 0 to 240 minutes for plasma glucose. | 0 to 240 minutes

SECONDARY OUTCOMES:
Plasma glucose concentrations | 0 to 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Amy Devitt-Maicher, PhD, Study Chair — Abbott Nutrition
Locations (1):
- Radiant Research, Cincinnati, Ohio, United States